CLINICAL TRIAL: NCT02169570
Title: Effect of Supplementary Vitamin D in Patients With Diabetes Mellitus and Pulmonary Tuberculosis (EVIDENT Study): a Randomized, Double Blind, Controlled Trial
Brief Title: Effect of Supplementary Vitamin D in Patients With Diabetes Mellitus and Pulmonary Tuberculosis
Acronym: EVIDENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Kashif Shafique, Assistant Professor/ Vice Dean SPH, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPH-P02
Record Dates: First submitted 2014-06-16; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes Mellitus; Pulmonary Tuberculosis
Keywords: Type 2 Diabetes Mellitus; Pulmonary Tuberculosis; Vitamin D; Calcium
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Tuberculosis, Pulmonary | interventions — Vitamin D; Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin D (Active Comparator): Vitamin D supplementation Anti Tuberculosis Treatment with 600,000 IU of (I/M) vitamin D3 for 3 doses at 0, 4 and 12 weeks and color and taste matched placebo for calcium for 3 months
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Placebo Calcium
- Placebo (Placebo Comparator): Anti Tuberculosis Treatment with placebo color matched for vitamin D and color and taste matched placebo for calcium
  Interventions: Dietary Supplement: Placebo Vit D; Dietary Supplement: Placebo Calcium
- Vitamin D and Calcium (Experimental): Vitamin D and Calcium supplementation Anti TuberculosisTreatment with 600,000 IU of (I/M) vitamin D3 for 3 doses at 0, 4 and 12 weeks with daily 1000 mg calcium carbonate for 3 months
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Other Names: Vitamin D3; cholecalciferol
  Arms: Vitamin D; Vitamin D and Calcium
Dietary Supplement: Calcium
  Arms: Vitamin D and Calcium
Dietary Supplement: Placebo Vit D
  Arms: Placebo
Dietary Supplement: Placebo Calcium
  Arms: Placebo; Vitamin D

SUMMARY:
Pakistan ranks fifth amongst high tuberculosis-(TB) burden countries, where TB persists as a major cause of misery and death. The Diabetes Mellitus-(DM) is also on rise in Pakistan and people suffering from DM are more prone to catch TB as compared to healthy individuals. This concurrence of two outbreaks may further increase the frequency of TB in Pakistan. The TB DM co-occurrence results in various clinical issues as TB in DM patient increases blood glucose, making DM more difficult to treat, while DM raises the risk of treatment failure, relapse and death among TB patients. In addition, both DM and TB usually coexist with micronutrients deficiencies like vitamin D, which has a vital role in immunity, insulin functioning and respiratory health. It has been suggested that the combined supplementation with vitamin D and calcium might be beneficial in improving the glucose metabolism but the current knowledge is very limited. In a resource restrained country with double burden of infectious and non-infectious diseases, an integrated approach with modification of treatment options may benefit in management of these outbreaks.

Therefore, this study aims whether vitamin D and calcium supplementation could influence the recovery in patients with TB of lung and DM.

DETAILED DESCRIPTION:
Pakistan is going through an epidemiological transition that subjects it to a dual burden of communicable and chronic diseases. According to WHO, Pakistan ranks seventh in diabetes prevalence and fifth amongst high TB burden countries. Pakistan faces challenges in controlling both these diseases with combine prevalence of 16%. This co-occurrence of DM and TB represents a big health risk in our population, as diabetes effects susceptibility to TB which makes more frequent treatment failure which could result in more community acquired TB infection. On the other hand, TB can worsen glycemic control in patients with diabetes. Moreover, overlapping of various drugs used in treatment might affect the glycemic control and pharmacokinetics of anti-TB treatment, resulting in the management of TB patients with DM more complex. Additionally, both DM and TB often coexist with micronutrients deficiencies like vitamin D and calcium. A vital role of vitamin D in immunity, insulin resistance and respiratory health has been suggested. Vitamin D and calcium deficiencies might adversely affect glycemic control, while combined supplementation with both of these micronutrients might be helpful in improving glucose metabolism which in turn will improve the treatment outcome for both these diseases. There is a suggestion that the combined supplementation with vitamin D and calcium might be beneficial in improving the glucose metabolism but the current knowledge is only limited to one randomized control trial in this co-morbid group carried out in India. Even in that trial independent effect of Vitamin D remain unknown as they used a combination therapy of calcium and vitamin D. Furthermore, that trial did not include radiological changes occurred during the follow-up period so that remains a major limitation. Therefore, this study will assess the role of supplementation with vitamin D and calcium in recovery (positive radiological changes, weight gain, sputum conversion, and glycemic control) of pulmonary TB patients with type 2 DM.The goal of our trial is to better understand the role of micro nutrients supplementation in among patients who have active TB and type 2 DM in their disease prognosis.

The objectives are as follows:

1. To determine the whether the 3 doses of vitamin D 600,000 IU at intervals of 4 weeks alone or in combination with calcium 1000mg for 3 months given with standard TB and type 2 DM treatment makes more rapid improvement in clinical indicators that are weight and TB score among 30 to 60 years old patients of active pulmonary TB with type 2 DM attending Ojha Institute of Chest Disease (OICD).
2. To determine the whether the mentioned doses of vitamin D and calcium with standard TB and type 2 DM treatments expedites radiological resolution and sputum conversion.
3. To determine whether the mentioned doses of vitamin D and calcium with standard TB and type 2 DM treatments is efficacious on glycemic control among these patients.
4. To guide future clinical treatment for such patients.

Methods:

Study Design and Setting:

A double blind randomized placebo-controlled trial at Ojha Institute of Chest Disease (OICD).

Duration of study: Three years after grant approval Sample size: We will require a sample size of 144 patients in each arm to measure an increase of ≥ 10% in weight gain and an improvement of 15% in chest radiograph among patients with combined supplementation of vitamin D and calcium as compared to placebo group. A total of 432 rounding off to 435 patients will be required to reject the null hypothesis at 5% level of significance with 80% power and 15% loss of follow up.

Sampling strategy:

We will approach all patients coming to OICD with diagnosed active pulmonary TB and type 2 DM, prior to commencement of anti-tuberculosis therapy (ATT). We will include both types of diabetic patients; either already diagnosed with type 2 DM or screened positive for type 2 DM after consenting for this study.

Total number of visits 7 (at 0, 4, 8, 12, 16, 24 weeks and 1 follow up)

Data collection Procedure Data will be collected by trained data collectors. Medical providers in the OICD OPDs would provide information about potential participants to data collectors, who would invite all patients initiating anti-TB treatment (ATT) to be considered enrolling in the study. On the basis of clinical history and records, and screening for type 2 DM, patients would be enrolled in this study. A block randomization; computer generated, stratified, random assignment list, would be used to randomize eligible participants. The patients in 3 study arms would either receive ATT with 600,000 IU of intramuscular (I/M) vitamin D3 (cholecalciferol) for 3 doses at 0, 4 and 12 weeks and color and taste matched placebo for calcium or ATT with 600,000 IU of (I/M) vitamin D3 for 3 doses at 0, 4 and 12 weeks with daily 1000 mg calcium carbonate or ATT with placebo color matched for vitamin D and color and taste matched placebo for calcium. All patients would be adjusted for oral hypoglycemic agents and insulin for glycemic control.

Chest radiographs, serum-25-(OH)D3 levels, serum calcium, Random Blood Sugar(RBS), Fasting Blood Sugar (FBS) and hemoglobin A1c (HbA1c) would be obtained at 0, 8, 16 and 24 weeks and sputum examination at 0, 4, 8, 12, 16 and 24 weeks of therapy. Clinical examination would be used to calculate a TB score for every visit. Weight would also be measured at all visits. At baseline other parameters including Complete Blood Count (CBC), Erythrocyte Sedimentation Rate (ESR), Liver Function Test (LFTs), lipid profile, serum albumin, and urine microalbumin would be tested. All blood test would be performed at Dow Diagnostic and Research Laboratory (DDRL) and Chest X-ray at Radiology department of DUHS Ojha campus. Consultant Radiologist will report on radiological finding and establishment of final diagnosis in outcome. Consultant Pulmonologist will select participant, follow up consultation, establishment of final diagnosis in outcome. All participants would be assured that no information regarding them would be shared to any one and that this information would be used only for research purpose. Pro forma, blood samples and chest x-ray would be marked by identification no. assigned to the participant. Data would be entered by data entry officer and then cleaned for any missing variables.

Data collection tools:

Pro forma would be used to collect basic demographic and clinical information. X-ray, sputum, blood and urine test from Radiology department of DUHS ojha campus and DDRL respectively.

Data analysis Plan:

Epi Data Entry software version 1.3 would be used for data entry. Data would be entered and cleaned for any missing entries. Data would be analyzed by 'intention-to-treat' analysis using software of SPSS version 16. Outcome variables would be reported by either by their means and standard deviations or percentages. Statistical comparisons at 0, 12 and 24 weeks would be performed using Pearson Chi-squared tests and Student's t-test for categorical and continuous variables respectively. A two-tailed p-value of < 0.05 would be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 60 years
* Patients having both TB and type 2 DM
* Patients consenting to participate
* No history of previous ATT
* Plane to have ATT and DM treatment

Exclusion Criteria:

* Age less than 30 years or greater than 60 years
* Pregnant women
* Patients having either TB or type 2 DM
* Patients refuse to participate
* Patients having extra-pulmonary TB or Multi-drug resistant MDR TB or relapse cases
* Patients having hepatic or renal diseases or HIV infection
* Patients having hypo- or hyper-parathyroidism
* Patients on corticosteroids or immunosuppressive or thiazides diuretics or any other drugs known to interfere with vitamin D levels

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 435 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | 0, 4, 8, 12, 16, 20 and 24 weeks and 6 months
  Weight will be measured by digital weighing machine.
Change in TB score | 0, 4, 8, 12, 16, 20 and 24 weeks, 6 months
  Clinical examination would be used to calculate it. It is a validated assessment tool developed to objectively measure change in the clinical status of TB patients. Its components include self-reported symptoms (cough, shortness of breath, night sweats, chest pain, haemoptysis), clinical signs (tachycardia, pallor, fever, auscultatory findings) body mass index (BMI) and mid-upper arm circumference (MUAC). The TB score so achieved could range from 0-13. TB scores would be divided in 3 severity classes; Severity Class I (TB score 0 to 5), Class II (TB score 6 - 7) and Class III (TB score ≥ 8).
Change Acid Fast Bacilli (AFB) smear (Sputum) | 0, 4, 8, 12, 16 and 24 weeks, 6 months
  Clearance of sputum
Change in chest X-ray | 0, 8, 16 and 24 weeks , 6 months
  Three separate methods of disease categorization would be used based on the classification of the National Tuberculosis and Respiratory Disease Association. This would include classification into 'minimally', 'moderately' and far advanced categories of radiographic infiltrates Secondly, cavity size ; No Cavity, Cavity size < 4 cm and ≥ 4 cm. Thirdly, the bilateral lung fields would be divided in to 3 zones (6 total) and disease extent would be recorded as 'Zone involvement' depending on active parenchymal and cavitary disease.

SECONDARY OUTCOMES:
Change Heamoglobin A1c (HbA1c) | 0, 8, 16 and 24 weeks, 6 months
  Blood test from Dow Diagnostic and Research Laboratory (DDRL). Blood sample will taken by phlebotomist for the HBA1c from the participants
Change in Fasting Blood Test (FBS) | 0, 8, 16 and 24 weeks, 6 months
  Blood test from Dow Diagnostic and Research Laboratory (DDRL). Blood sample will taken by phlebotomist for the FBS from the participants after 8-10 hours of fasting
Change in Random Blood Sugar (RBS) | 0, 8, 16 and 24 weeks, 6 months
  Blood test from Dow Diagnostic and Research Laboratory (DDRL). Blood sample will taken by phlebotomist for the RBS from the participants

CONTACTS AND LOCATIONS:
Overall Officials: Kashif - Shafique, PhD, Principal Investigator — School of Public Health, Dow University of Health Sciences, Karachi, Pakistan
Locations (1):
- School of Public Health, Dow university of Health Sciences, Karachi, Sindh, Pakistan